CLINICAL TRIAL: NCT04108689
Title: Internet-based Acceptance and Commitment Training for Elite Ice Hockey Players: an Open-trial
Brief Title: Internet-based Acceptance and Commitment Training for Elite Ice Hockey Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tobias Lundgren, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-ACT-Hockey
Record Dates: First submitted 2019-09-23; First posted 2019-09-30 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Performance Enhancement; Performance Anxiety; Mental Health
Keywords: internet intervention; applied sport psychology; performance enhancement; acceptance and commitment training; elite ice hockey
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- I-ACT (Experimental): I-ACT is short for Internet-Acceptance and Commitment Training
  Interventions: Behavioral: I-ACT

INTERVENTIONS:
Behavioral: I-ACT — An internet-based behavioral psychotherapy intervention to enhance athletic performance in elite ice hockey players.

SUMMARY:
The aim of this study is to investigate whether an internet-based psychological training program will enhance performance and affect mental health related factors in elite ice hockey players. The psychological training program is based on Acceptance and Commitment Therapy (ACT), a modern form of Cognitive Behavior Therapy, and is delivered over the internet (hence called "I-ACT"). Elite players in Sweden will be invited before the 2019/2020 season. I-ACT will start for enrolled participants during the first week of October 2019 (30th September- 2nd October depending on the schedule of the particular league; approximately 5 games have then been played in the leagues eligible for participation). I-ACT consists of seven weekly modules/chapters with ACT content and participants also have a psychological trainer in the program that they can contact via a chat function on the web platform. Participants will have completed I-ACT the 17th of November 2019. When I-ACT starts in October, other eligible players will have the opportunity to leave their notice of interest for participation in the study and to take part of I-ACT in a later stage of the season. This concurrent "waiting list" is not a waiting list control group in any sense. It only gives further eligible players the opportunity to enroll in the study for a consecutive start of the psychological training program. I-ACT will start for this second group of players during the last week in november (25th November 2019), and finish I-ACT the 12th January 2020. These two consecutive groups of I-ACT participants will be considered the experimental group. However, due to the length of the ice hockey season the second group will only have follow-up measurements at 1 month for female players (the women's league ends in February 2020) and 2 months for male players (the men's leagues ends in March 2020). Official statistics will be collected from the leagues and enrolled participants will be compared to non-participant players in the leagues to compare the effectiveness of I-ACT on ice hockey performance. Only within-group comparisons will be made for secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Playing ice hockey on elite level in any of the following leagues: Svenska damhockeyligan (SDHL, the Swedish premier ice hockey league for women), Svenska hockeyligan (SHL, the Swedish premier ice hockey league for men), Hockeyallsvenskan (the Swedish second highest league in ice hockey for men).

Exclusion Criteria:

* Players currently participating in any other individual psychological training program.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Objective ice hockey performance data: goals | Pre (aggr. to a single score from 5 games pre),during(aggr. to single scores from 5 game intervals until end of interv),post(aggr. to a single score from 5 games post), followup(aggr. to single scores from 5 game intervals up to 4-16 weeks = season ends)
  Scored goals by a player. Data is always aggregated from a 5 game interval into a single score. The statistics will be collected by the official statistic systems for eligible leagues, which in turn will be used in the study.
Objective ice hockey performance data: assists | Pre (aggr. to a single score from 5 games pre),during(aggr. to single scores from 5 game intervals until end of interv),post(aggr. to a single score from 5 games post), followup(aggr. to single scores from 5 game intervals up to 4-16 weeks = season ends)
  Made assists by a player. Data is always aggregated from a 5 game interval into a single score. The statistics will be collected by the official statistic systems for eligible leagues, which in turn will be used in the study.
Objective ice hockey performance data: total points | Pre (aggr. to a single score from 5 games pre),during(aggr. to single scores from 5 game intervals until end of interv),post(aggr. to a single score from 5 games post), followup(aggr. to single scores from 5 game intervals up to 4-16 weeks = season ends)
  Total points by a player (number of goals + assists). Data is always aggregated from a 5 game interval into a single score. The statistics will be collected by the official statistic systems for eligible leagues, which in turn will be used in the study.
Objective ice hockey performance data: +/- statistics | Pre (aggr. to a single score from 5 games pre),during(aggr. to single scores from 5 game intervals until end of interv),post(aggr. to a single score from 5 games post), followup(aggr. to single scores from 5 game intervals up to 4-16 weeks = season ends)
  +/- statistics for a player (number of goals scored and conceded by a team while a certain player is on the ice) . Data is always aggregated from a 5 game interval into a single score. The statistics will be collected by the official statistic systems for eligible leagues, which in turn will be used in the study.
Objective ice hockey performance data: saving percent (only for goalkeepers) | Pre (aggr. to a single score from 5 games pre),during(aggr. to single scores from 5 game intervals until end of interv),post(aggr. to a single score from 5 games post), followup(aggr. to single scores from 5 game intervals up to 4-16 weeks = season ends)
  Saving percent (only for goalkeepers). Data is always aggregated from a 5 game interval into a single score. The statistics will be collected by the official statistic systems for eligible leagues, which in turn will be used in the study.

SECONDARY OUTCOMES:
The Values, Acceptance and Mindfulness Scale for Ice Hockey (VAMS) | Pre-intervention, during(every week for the 7 week interv), post-intervention, and follow up at every 4th week until end of season (up to 4-16 weeks depending on the participants league and if the player is enrolled in the first or second start of I-ACT)
  Measures behavioral and psychological flexibility in ice hockey. 11 items. Total range is 11-77. A high value represent a better outcome. Three subscales; Acceptance (5 items, points range 1-35); Values (3 items, points range 1-21); Mindfulness (3 items, points range 1-21). The subscale scores are summed for total score.
Subjective performance | Pre-intervention, during(every week for the 7 week interv), post-intervention, and follow up at every 4th week until end of season (up to 4-16 weeks depending on the participants league and if the player is enrolled in the first or second start of I-ACT)
  Players subjective rating of performance. This is a single-item measure developed for this study asking players to rate their own hockey performance during the last week on a scale of 1-10 (1 = extremely poor, 10 = extremely good).
Brunnsviken Brief Quality of Life Scale (BBQ) | Pre-intervention, during intervention (at week 4), post-intervention, and follow up at every 4th week until end of season (up to 4-16 weeks depending on the participants league and if the player is enrolled in the first or second start of I-ACT)
  Measures quality of life. 12 items. Total range is 0-96. A higher value is the better outcome.
Insomnia Severity Index (ISI) | Pre-intervention, during intervention (at week 4), post-intervention, and follow up at every 4th week until end of season (up to 4-16 weeks depending on the participants league and if the player is enrolled in the first or second start of I-ACT)
  Measures sleep impairment and quality
General Anxiety Disorder 7-item Scale | Pre-intervention, post-intervention, and follow up at every 4th week until end of season (up to 4-16 weeks depending on the participants league and if the player is enrolled in the first or second start of I-ACT)
  Measures generalised anxiety. 7 items. Total range is 0-21. A low value is the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Lundgren, PhD, Principal Investigator — Centre for Psychiatry Research, Department of Clinical Neuroscience, Karolinska Institutet
Locations (1):
- Centre for Psychiatry Research, Department of Clinical Neuroscience, Karolinska Institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No